CLINICAL TRIAL: NCT01032122
Title: Efficacy and Safety of Rituximab, an Anti-CD20 (Cluster of Differentiation Antigen 20) Therapeutic Agent, in Metastatic Melanoma: a Pilot Study
Brief Title: Rituximab in Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the only reason is that recruitment was not sufficient to meet the planned patient numbers, because complete remissions are still infrequent.
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stephan N. Wagner, MD, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIMM1
Record Dates: First submitted 2009-09-19; First posted 2009-12-15 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; rituximab; metastatic; stage IIIc/IV; stem cell; overall survival; disease free interval; anti-CD20 therapy
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab (Experimental)
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — induction phase: 375mg/m² qw, 4wks; followed by maintenance phase: 375mg/m², every 8 wks; duration: 2 years.
  Other Names: mabthera; rituxan

SUMMARY:
The purpose of this study is to determine whether rituximab as an adjuvant therapy in clinical stage IIIc / IV (no evidence of disease, AJCC (American Joint Committee on Cancer) 2002) melanoma patients is safe and prolongs overall survival and disease-free interval.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified non-ocular melanoma stage IIIc/IV, no evidence of disease

Exclusion Criteria:

* ECOG (Eastern Cooperative Oncology Group) performance status > 2
* Ocular melanoma
* Immunodeficiency syndromes or hypogammaglobulinaemia
* Active autoimmune diseases
* Treatment with immunosuppressive agents other than steroids
* Depressed bone marrow function (Leukopenia <3000, platelet count <100.000)
* Cardiac insufficiency NYHA (New York Heart Association) IV
* active Hepatitis B,C, or HIV infection
* Pregnancy or lactation
* Interstitial pulmonary disease
* Former treatment with anti-CD20 antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
disease-free interval | 42 months

SECONDARY OUTCOMES:
overall survival | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wagner, MD, Principal Investigator — Med Univ Vienna; Alice Pinc, MD, Principal Investigator — Medical Univ Vienna
Locations (1):
- General Hospital Vienna, Dep. of Dermatology, Division of Immunology and Infectious Diseases, Vienna, Austria